CLINICAL TRIAL: NCT05750953
Title: Project Title: Nurse Assisted eHealth Service From Hospital to Home: Ameliorating Burden of Treatment Among Patients With Non-Communicable Diseases
Brief Title: Nurse-assisted Intervention "eHealth@ Hospital -2-home"
Acronym: Ehealth@H2H
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stavanger (Other)
Collaborators: Helse Stavanger HF (Other Government); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 301472
Record Dates: First submitted 2022-11-02; First posted 2023-03-02 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-12

CONDITIONS: Non Communicable Diseases; Heart Failure; Colon Rectal Cancer
MeSH Terms: conditions — Noncommunicable Diseases; Heart Failure; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with intervention and control group
Who Masked: Investigator
Masking Description: Randomization will be blinded for the study statistician and researchers performing the data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eHealth@H-2-H (Experimental): The intervention group will participate in a 42-day nurse-assisted RPM intervention "eHealth@ Hospital-2-Home". The intervention includes monitoring of vital signs, self-reports of symptoms, health and well-being, access to information about illness and health resources , and communication between the patients and a hospital-based Nurse Navigator.
  Interventions: Behavioral: eHealth@Hospital-2-Home
- Care as usual (No Intervention): The control group will receive care as usual

INTERVENTIONS:
Behavioral: eHealth@Hospital-2-Home — At hospital discharge, the intervention group will receive a wireless, portable personal computer system (i.e., IPAD) that includes the eHealth application MyDignio supplied by a certified m-Health company. MyDignio app is linked to monitoring devices by Bluetooth for each patient to daily and weekly measure clinical measures such as blood pressure, pulse, temperature, and weight, and self-reported symptoms and well-being, and daily report clinical measurements to the Nurse Navigators employed in the two hospitals. The patients will receive training from the nurses on how to log on and use the MyDignio app and the monitoring devices. Telephone contact details including information about how to access technical support will be provided to each study participant shortly following discharge.
  Other Names: nurse-assisted eHealth intervention on self-management among patients with Non-Communicable Disease
  Arms: eHealth@H-2-H

SUMMARY:
A randomized controlled trial with non-communicable disease patients from two medical hospitals in Norway will be recruited prior to hospital discharge. The intervention group will participate in a 42-day nurse-assisted eHealth intervention "eHealth@ Hospital-2-Home". The intervention includes monitoring the patient's vital signs, self-reports of symptoms, health and well-being, communication between the patients and a Nurse Navigator in the hospital, and access to information about illness and health resources.

DETAILED DESCRIPTION:
Heart failure (HF) and colon-rectal cancer (CRC) are two non-communicable diseases (NCDs) prone to a high rate of hospital admissions and re-admissions, and complex health care needs. For many patients with HF and CRC, self-management following hospitalization can be a challenge, and they may leave the hospital unprepared for self-managing their disease at home. The randomized controlled trial with NCD patients from two medical hospitals in Norway. Patients will be recruited before hospital discharge. The intervention group will participate in a 42-day nurse-assisted remote patient monitoring (RPM) intervention "eHealth@ Hospital-2-Home". The RPM intervention includes monitoring of patients' vital signs, self-reports of symptoms, health and well-being, communication between the patients and a Nurse Navigator in the hospital, and access to information about illness and health resources. The control group will receive care as usual. Data collection will take place before the intervention (baseline), at the end of the intervention (post-1), and 6 months after baseline (post-2). Data will be according to intention to treat principles. Qualitative data will be analyzed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* All participants: symptomatic HF or surgically treated for either colon or rectal cancer (Colon-Rectal Cancer Duke's class 1-3, curative), able to speak and write Norwegian

Exclusion Criteria:

* Heart failure population: patient is on a waiting list for a heart transplant, requires a Left Assist Ventricular Device (LVAD), and has a life expectancy <6 months
* Colon-rectal cancer population: metastatic cancer, Surgical Complication Score > 3, and acute medical crisis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient confidence in self-management activities. | Baseline (at discharge), post-1 (42 days following baseline, at the end of the intervention), and post-2 (6 months after baseline)
  Change in the patient's confidence in self-management of heart failure or colon-rectal cancer disease between baseline and post-1 and 2 will be measured by the 6 items questionnaire Self-Efficacy for Managing Chronic Disease". Values: 1-10. A higher score mean a better outcome.

SECONDARY OUTCOMES:
Change in patient experience with treatment and self-management. | Baseline (at discharge), post-1(42 days following baseline, at the end of the intervention) , and post-2 (6 months after baseline)
  Change in the patient's experience with treatment and self-management of heart failure and colon-rectal cancer between baseline and post-1 and 2 will be measured by the questionnaire "Patient Experience with Treatment and Self-management" with four dimensions of Medical information (Values:1-6); Monitoring health (Values: 1-6); Medications (Values 1- 5); Medical appointments (Values: 1-5). Higher scores means a worse outcome.
Change in patient experience of health condition and how it affects daily life. | Baseline (at discharge), post-1 (42 days following baseline, at the end of the intervention), and post-2 (6 months after baseline)
  Change in the patient's Health Related Quality of Life between baseline and post 1 and 2 will be measured with the European Quality of life 5 Dimensions -5 Levels questionnaire. Values: 1-5, were higher scores mean worse outcome, and on a visual analog scale from 0-100, were higher scores mean better outcome.
Change in patient experience of constructive support from healthcare personnel | Baseline (at discharge), post-1 (42 days following baseline, at the end of the intervention), and post-2 (6 months after baseline)
  Change in perceived support between baseline and post-1 and 2 will be measured using 12 items on constructive support. Values: 1-5-point. Higher score mean worse outcome.
Change in patient experience of shared decision-making. | Baseline (at discharge), post-1 (42 days following baseline, at the end of the intervention), and post-2 (6 months after baseline)
  Change in the patient's experience of shared decision-making between baseline and post-1 and 2 will be measured using the 3 items questionnaire "CollaboRATE" Value: 0-10. Higher score mean better outcome.
Change in health care utilization | Baseline (at discharge), post-1 (42 days following baseline, at the end of the intervention), and post-2 (6 months after baseline)
  Change in health care utilization between baseline and post-1 and 2 will be measured using patients' self-reports of number of visits to the primary healthcare service (i.e., General Practitioner, municipal emergency department) and/or the specialist healthcare service (i.e., outpatient clinic). Fewer visits mean better outcome.
Days alive and out of hospital | Post-2 (6 months after baseline)
  Days alive and out of hospital (Cohn 2009) will be collected from hospital records and subtracting the number of days spent away from home due to hospitalisation from the date of discharge up to date of death/six months (Post-2), i.e. possible range will be 0-180 days.
Time to first readmission or death | Time of first readmission within six months or death
  Time of first readmission within six months will be collected from hospital records, as will date of death (dod) for those who died within six months from the date of discharge from the primary hospitalisation. The first of these dates will define the endpoint for this outcome.

OTHER OUTCOMES:
Patient satisfaction with using the technology. | Post-1 (42 days following baseline, at the end of the intervention)
  Patient satisfaction with using the technology will be measured by the Post-Study System Usability Questionnaire. Values: 1-7. Higher score mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Husebø, PhD, Principal Investigator — University of Stavanger; Ingvild M Morken, PhD, Principal Investigator — University of Stavanger; Marianne Storm, PhD, Principal Investigator — University of Stavanger
Locations (1):
- Anne Marie Lunde Husebø, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No
According to legal and ethical legislation and approvals.